CLINICAL TRIAL: NCT07272486
Title: Effect of Virtual Reality and Classical Music Therapy on Blood Pressure and Anxiety in Patients With Hypertensive Urgency
Brief Title: The Use of Virtual Reality and Music Therapy for Hypertensive Urgency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, Associate Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-24-7802; E2-24-7802 (Other: Ankara Bilkent City Hospital)
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypertensive Urgency; Primary Hypertension
Keywords: Hypertensive Urgency; Primary Hypertension; Virtual Reality Therapy; Classical Music Therapy; Stress Reduction; Blood Pressure Control; Emergency Department
MeSH Terms: conditions — Hypertensive Crisis; Essential Hypertension; Emergencies | interventions — Captopril

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm parallel assignment model in which participants are randomized in a 1:1 ratio to receive either standard pharmacological treatment alone or standard treatment combined with virtual reality and classical music therapy. All interventions are delivered concurrently with routine management in a controlled emergency department environment, and participants are followed for 240 minutes with repeated blood pressure and anxiety assessments
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Pharmacological Treatment (Active Comparator): Participants in this arm will receive standard oral antihypertensive treatment consisting of 25 mg captopril. Additional doses (25 mg at 30 minutes and 25 mg at 60 minutes, total 75 mg) will be administered if MAP reduction of ≥25% is not achieved. Rescue therapy with IV nitrate (0.1 mg/kg/min) will be used if blood pressure remains uncontrolled after 90 minutes, following routine emergency department protocol. No VR or music therapy is administered in this arm.
  Interventions: Drug: Captopril 25Mg Tab
- Standard Treatment + VR and Classical Music Therapy (Experimental): Participants in this arm will receive standard oral antihypertensive treatment (25 mg captopril; additional doses at 30 and 60 minutes if needed) combined with virtual reality exposure and classical music therapy. Patients will view a calming VR environment of their choice for approximately 20 minutes while listening to a selected classical music piece. VR and music therapy are administered concurrently in a quiet and dimly lit room. Rescue therapy with IV nitrate will be used according to the same emergency department protocol as the control group.
  Interventions: Drug: Captopril 25Mg Tab; Device: Virtual Reality Exposure; Behavioral: Classic Music Therapy

INTERVENTIONS:
Drug: Captopril 25Mg Tab — This drug is administered to participants in both study arms. Standard oral antihypertensive treatment with 25 mg captopril is given at baseline. Additional 25 mg doses may be administered at 30 and 60 minutes if ≥25% MAP reduction is not achieved. Rescue therapy with IV nitrate may be used after 90 minutes according to routine emergency department protocol
Device: Virtual Reality Exposure — This intervention is administered only to participants in the 'Standard Treatment + VR and Classical Music Therapy' arm. Participants view a calming virtual environment of their choice for approximately 20 minutes using a non-proprietary VR headset. The session is delivered concurrently with standard antihypertensive treatment in a quiet, dimly lit room
  Arms: Standard Treatment + VR and Classical Music Therapy
Behavioral: Classic Music Therapy — This intervention is administered only to participants in the 'Standard Treatment + VR and Classical Music Therapy' arm. Participants listen to one of several selected classical music pieces at a comfortable volume (40-60 dB) during the VR exposure. Music therapy is applied simultaneously with standard antihypertensive treatment to support relaxation.
  Arms: Standard Treatment + VR and Classical Music Therapy

SUMMARY:
This study aims to evaluate whether virtual reality (VR) and classical music therapy, when added to standard antihypertensive treatment, can improve blood pressure control and reduce anxiety in patients presenting to the emergency department with hypertensive urgency. Patients with primary hypertension and no signs of end-organ damage will be randomly assigned to receive either standard treatment alone or standard treatment combined with VR and classical music. Blood pressure will be monitored at multiple time points over a 240-minute period, and anxiety will be assessed using the State Anxiety Inventory (STAI-I). The study seeks to determine if these non-pharmacological interventions can enhance the effectiveness of routine management of hypertensive urgency.

DETAILED DESCRIPTION:
Hypertensive urgency is characterized by severely elevated blood pressure without evidence of acute target-organ damage. Standard management typically involves the gradual reduction of blood pressure using oral antihypertensive agents such as captopril. Emotional stress and anxiety can contribute to elevated sympathetic activity, potentially worsening blood pressure control. Virtual reality (VR) environments and classical music therapy have been shown in prior studies to reduce stress, improve patient comfort, and modulate physiological responses.

In this randomized controlled study, patients with primary hypertension who present to the emergency department with hypertensive urgency will be assigned to one of two groups: standard pharmacological treatment alone or standard treatment combined with VR exposure and classical music therapy. The intervention will be delivered in a quiet and dimly lit room, and blood pressure will be measured at predefined intervals over 240 minutes. Anxiety levels will be assessed at baseline and at the end of the monitoring period using the State Anxiety Inventory (STAI-I).

This study aims to determine whether VR and classical music can enhance routine management by improving blood pressure reduction and decreasing anxiety levels during acute hypertensive episodes. Findings may support the incorporation of non-pharmacological strategies into the emergency management of hypertensive urgency.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of primary hypertension
* Presentation to the emergency department with hypertensive urgency
* Absence of any signs of acute end-organ damage
* Ability to understand the study and provide informed consent
* Able to cooperate with serial blood pressure measurements

Exclusion Criteria:

* Age younger than 18 years
* Diagnosis of secondary hypertension
* Any medication intolerance or known hypersensitivity to captopril or nitrate therapy
* Current severe psychiatric disorder or cognitive impairment interfering with participation
* Contraindications to using virtual reality (history of severe vertigo, epilepsy, motion sickness, etc.)
* Hemodynamic instability requiring immediate high-intensity medical intervention
* Pregnancy or breastfeeding
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Mean Arterial Pressure (MAP) at 30 Minutes | Baseline (after 10 minutes of rest) and 30 minutes after treatment initiation
  Mean arterial pressure will be measured at baseline (after 10 minutes of rest) and again at 30 minutes after the initial treatment. The primary endpoint is the percentage reduction in MAP at 30 minutes compared with baseline, with a target reduction of at least 25%.

SECONDARY OUTCOMES:
Change in State Anxiety Level (State Anxiety Inventory - Form I) | Baseline and 240 minutes
  State anxiety will be measured using the State Anxiety Inventory - Form I (STAI-I), a validated 20-item scale assessing situational anxiety. Total scores range from 20 to 80, with higher scores indicating higher levels of state anxiety. STAI-I will be administered at baseline and at 240 minutes to evaluate changes during the observation period.
Incidence of Adverse Events | Up to 240 minutes
  Frequency and type of adverse events related to antihypertensive medication or VR/music therapy (e.g., dizziness, nausea, hypotension) will be documented during the entire observation period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vorwerg-Gall S, Stamm O, Haink M. Virtual reality exergame in older patients with hypertension: a preliminary study to determine load intensity and blood pressure. BMC Geriatr. 2023 Aug 30;23(1):527. doi: 10.1186/s12877-023-04245-x. PMID 37644380
- [Result] Jiravska Godula B, Jiravsky O, Matheislova G, Kuriskova V, Valkova A, Puskasova K, Dokoupil M, Dvorakova V, Prifti A, Foral D, Jiravsky F, Hecko J, Hudec M, Neuwirth R, Miklik R. Virtual Reality for Patient Education about Hypertension: A Randomized Pilot Study. J Cardiovasc Dev Dis. 2023 Nov 29;10(12):481. doi: 10.3390/jcdd10120481. PMID 38132649
- [Result] Patel KK, Young L, Howell EH, Hu B, Rutecki G, Thomas G, Rothberg MB. Characteristics and Outcomes of Patients Presenting With Hypertensive Urgency in the Office Setting. JAMA Intern Med. 2016 Jul 1;176(7):981-8. doi: 10.1001/jamainternmed.2016.1509. PMID 27294333
- [Result] Kulkarni S, Glover M, Kapil V, Abrams SML, Partridge S, McCormack T, Sever P, Delles C, Wilkinson IB. Management of hypertensive crisis: British and Irish Hypertension Society Position document. J Hum Hypertens. 2023 Oct;37(10):863-879. doi: 10.1038/s41371-022-00776-9. Epub 2022 Nov 22. PMID 36418425
- [Result] Qin Z, Zhou C, Zhu Y, Wang Y, Cao H, Li W, Huang Z. Virtual Reality for Hypertension in Tooth Extraction: A Randomized Trial. J Dent Res. 2022 Apr;101(4):400-406. doi: 10.1177/00220345211049393. Epub 2021 Nov 26. PMID 34825613
- [Result] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension global hypertension practice guidelines. J Hypertens. 2020 Jun;38(6):982-1004. doi: 10.1097/HJH.0000000000002453. No abstract available. PMID 32371787